CLINICAL TRIAL: NCT03633162
Title: Maternal Grandmothers in the Born in Guangzhou Cohort Study
Acronym: MGBIG
Status: Recruiting | Type: Observational
Sponsor: Guangzhou Women and Children's Medical Center (Other)
Collaborators: Children's Hospital Medical Center, Cincinnati (Other); University of Birmingham (Other)
Responsible Party: Principal Investigator, Xiu Qiu, Director of the Born in Guangzhou Cohort Study, Guangzhou Women and Children's Medical Center
Other Study IDs: 2018041801; 81673181 (Other Grant/Funding Number: National Natural Science Foundation of China); 201508030037 (Other Grant/Funding Number: Guangzhou Science and Technology Bureau, Guangzhou, China)
Record Dates: First submitted 2018-07-23; First posted 2018-08-16 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Hereditary Transmission; Immune Development; Childhood Obesity; Host and Microbiome; Neurodevelopment
Keywords: Maternal Grandmother; Genes; Immune; Cohort; Child development
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — blood, buccal mucosal cells, stool, urine, fingernail and hair
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other:

SUMMARY:
The MGBIG is a study exploring cross-generational effects in 5000 women and their children and grandchildren located in Guangzhou, China. Its initial aim is to facilitate research on understanding the interplay between genes and environmental factors on disease etiology and on explaining the cause of the disease from the perspective of "grandmother-mother-child" heredity. Data are collected regarding environmental exposures, lifestyle, and social support on grandmother from birth to old age. Biological samples including blood and tissue samples are collected.

DETAILED DESCRIPTION:
It was previously believed that heredity strictly follows Mendel's laws, but recent studies have found that through placental material exchange, mammals may transfer maternal immune-related factors vertically, thus promoting the protection of "non-heredited maternal antigenic traits". Thus, the transmission of reproductive information across generations is realized. Since the unusual genetic pattern of the X chromosome, grandmother's influence may be gender specific. Since grandchildren were usually took care by grandparents in China, it could be achievable to attach and recruit maternal grandmother together with mother and children. Cohort including three generations of women is rare in Asia at present. In the MGBIG, extensive information including demographic characteristics, lifestyle, history of diseases, mental health, and behaviors is collected from the participants. Longitudinal follow up and surveillance of common chronic diseases are also to be conducted. The MGBIG intends to recruit maternal grandmothers to study the effects of maternal genetic and environmental exposure on the health of their children and grandchildren.

ELIGIBILITY:
Inclusion Criteria:

1. Maternal Grandmother' grandchildren delivered in Guangzhou Women and Children's Medical Center
2. Baseline information of maternal grandmother's daughter during pregnancy available

Exclusion Criteria:

1. Significant cardiovascular abnormalities
2. Intelligent obstacle, intellectual disabilities or gawkish condition

Ages: 36 Years to 100 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — female
Study Population: All maternal grandmothers of the children in the Born in Guangzhou Cohort Study (BIGCS) would be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2018-05-21 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2038-12-31 (Estimated)

PRIMARY OUTCOMES:
Haplotypes transfered by non-inherited maternal antigens from maternal grandmother to female offspring | From the date of her daughter get pregnant until the date her grandchild/grandchildren is/are given birth
  Assessed by analyses of MHC haplotypes, HLA haplotypes, and levels of non-inherited maternal antigens of mother and offspring, and pregnancy complication of maternal grandmothers and mothers

SECONDARY OUTCOMES:
Serum levels of Inflammatory factors at grandchildren's birth and early neonatal life | At the birth date of her grandchild/grandchildren, at the date 42 days after the birth of the certain grandchild/grandchildren
  Assessed by analyses of IL-1, IL-6, IL-10, IL-12, etc.
The prevalence of eczema of grandchildren | At the age of 6 weeks, 6 months, 1year, 3 years, 6 years, 12years and 18years of grandchildren
  Assessed by self-reported time of onset and electronic medical record
The incidence of asthma of grandchildren | At the age of 6 months, 1year, 3 years, 6 years, 12years and 18years of grandchildren
  Assessed by self-reported time of onset and electronic medical record
The prevalence of Allergic rhinitis of grandchildren | At the age of 6 months, 1year, 3 years, 6 years, 12years and 18years of grandchildren
  Assessed by self-reported time of onset and electronic medical record
The prevalence of Food allergy of children and grandchildren | At the age of 6 months, 1year, 3 years, 6 years, 12years and 18years of grandchildren
  Assessed by self-reported time of onset and electronic medical record
Changes of body composition of grandchildren | At age of 3 years,6 years, 12years and 18years
  Body composition is assessed using Dual Energy X-Ray Absorptiometry
Changes of bone density of grandchildren | At age of 3 years,6 years, 12years and 18years
  Bone density is assessed using Dual Energy X-Ray Absorptiometry

CONTACTS AND LOCATIONS:
Overall Officials: Xiu Qiu, PhD, Principal Investigator — Guangzhou Women and Children's Medical Center, China
Locations (1):
- Guangzhou Women and Children's Medical Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Qiu X, Lu JH, He JR, Lam KH, Shen SY, Guo Y, Kuang YS, Yuan MY, Qiu L, Chen NN, Lu MS, Li WD, Xing YF, Zhou FJ, Bartington S, Cheng KK, Xia HM. The Born in Guangzhou Cohort Study (BIGCS). Eur J Epidemiol. 2017 Apr;32(4):337-346. doi: 10.1007/s10654-017-0239-x. Epub 2017 Mar 20. PMID 28321694
- [Background] Kinder JM, Jiang TT, Ertelt JM, Xin L, Strong BS, Shaaban AF, Way SS. Cross-Generational Reproductive Fitness Enforced by Microchimeric Maternal Cells. Cell. 2015 Jul 30;162(3):505-15. doi: 10.1016/j.cell.2015.07.006. Epub 2015 Jul 23. PMID 26213383